CLINICAL TRIAL: NCT04383262
Title: A 12-Week Randomized, Double-Blind, Placebo-Controlled Clinical Trial to Assess the Efficacy of Oral Fosamprenavir for Laryngopharyngeal Reflux
Brief Title: Fosamprenavir for Laryngopharyngeal Upper Airway Tissue Treatment and Enzyme Reduction
Acronym: FLUTTER
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Nikki Johnston, Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO00056069
Record Dates: First submitted 2020-05-01; First posted 2020-05-12 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Laryngopharyngeal Reflux
MeSH Terms: conditions — Laryngopharyngeal Reflux | interventions — fosamprenavir

STUDY DESIGN:
Intervention Model Description: Proof-of-Concept Efficacy Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: We have partnered with Froedtert Hospital's Investigative Drug Services in order to randomize subjects to either treatment or placebo. Only FH IDS will have the key linking subjects to treatment groups, and the power to conduct an emergency unblinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oral Fosamprenavir pills (Experimental): FOS: 1,400 mg fosamprenavir calcium b.i.d. (AM/PM) for 12 weeks
  Interventions: Drug: Fosamprenavir Calcium
- Placebo (Placebo Comparator): Sodium Alginate: for 12 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Fosamprenavir Calcium — A repurposing approach, prospective, placebo-controlled clinical trial of FOS-SA (used at 1,400 mg fosamprenavir calcium, twice daily) for 12 weeks in medically refractory patients with clinically diagnosed moderate/severe LPR (RSI > 13, RFS > 7 and MII-pH confirmed laryngeal reflux event[s]).
  Arms: Oral Fosamprenavir pills
Other: Placebo — Non-active placebo pill formulation
  Arms: Placebo

SUMMARY:
Laryngopharyngeal Reflux (LPR) is a common condition that causes symptoms like chronic cough, throat clearing, hoarseness, and trouble swallowing. If not treated, LPR can lead to long-term throat damage and may increase the risk of throat cancer. More than 20% of the people in the United States are estimated to have LPR, yet there is no effective medication approved to treat it. Drugs called proton pump inhibitors (PPIs) are often used to treat LPR, even though they were designed for stomach acid problems. These medications reduce acid but do not stop reflux from happening, so they often do not help LPR patients. Despite poor results, PPIs are widely prescribed, are very costly, and can cause side effects.

Research shows that a digestive enzyme called pepsin plays a key role in LPR. Pepsin can damage the throat and voice box even when acid is not present. Laboratory studies found that certain HIV medications can block damage caused by pepsin. People taking these medications for HIV appear to have a much lower rate of LPR. This study will test fosamprenavir, an FDA-approved HIV drug, as a treatment for LPR. We will conduct a 14-week, double-blind, placebo-controlled clinical trial in patients with LPR who did not improve with standard treatment. Participants will receive either fosamprenavir or placebo, randomly, and symptoms will be measured before and after treatment using standard questionnaires and daily symptom tracking.

Because there is no effective medical treatment for LPR. this study aims to test a safe, existing drug that targets the underlying cause of the disease.

DETAILED DESCRIPTION:
Laryngopharyngeal reflux (LPR) causes chronic cough, throat clearing, hoarseness, and dysphagia and if left untreated can promote the development of laryngeal cancer. More than 20% of the United Stated population suffer from LPR, yet there is no effective medical therapy. Proton pump inhibitors (PPIs), which inhibit gastric acid production but do not prevent reflux events, continue to be prescribed for LPR despite their poor efficacy for this patient population, high cost ($26 billion/year), and associated risks. Pepsin, detected in the airway of these patients and now known to cause laryngeal inflammation and promote disease independent of gastric acid, is a key therapeutic target. We report preclinical studies of select HIV inhibitors that bind to and inhibit pepsin and thus hold promise for the treatment of LPR. In support, a very low incidence of LPR was found in patients taking these drugs compared to the general population. HIV inhibitors are ideal drugs to repurpose because they target a foreign virus. Thus, a repurposing approach can be used to safely perform proof of concept testing of the efficacy of a pepsin inhibitor for LPR.

The objective of this study is to evaluate the efficacy and safety of fosamprenavir (FOS), administered orally for improving symptoms of laryngopharyngeal reflux (LPR). The Specific Aim of this project is to perform a 12-week randomized, double-blind, placebo-controlled clinical trial to assess the efficacy of fosamprenavir pills for LPR. Fosamprenavir will be used at the FDA approved, manufacturers recommended dose for HIV for 12 weeks in medically refractory patients with clinically diagnosed moderate/severe LPR and combined multi-channel intraluminal impedance - pH (MII-pH) confirmed laryngeal reflux events. Routine clinical outcome measures for LPR (Reflux Symptom Index, Reflux Finding Score, Voice Handicap Index) will be documented pre- and post-treatment with Oral Fosamprenavir for LPR (n = 52) and placebo (n = 52). Additional research measures will include repeat administration of a newly created Daily Symptom Reflex Diary, as well as an intermittently distributed Patient Global Impression - Static & Change scales.

ELIGIBILITY:
1. Clinical diagnosis of LPR 2. Age ≥ 18 years 3. RSI > 13 4. RFS > 7 5. Documented LPR by MII-pH testing (> 1 proximal event) 6. Failed 3 month bid PPI therapy 7. Attending laryngology clinic with study providers, and having flexible laryngoscopy and MII-pH testing per routine clinical care with a minimum of three months between clinic visits (standard practice) 8. For continued participation after ATRU V1/V2:

1. Hepatic Function Panel must be within normal limits
2. Results from V1 safety labs must all be within normal limits
3. Patient agrees not to make any changes to their usual diet and/or anti-reflux medications during the study.
4. Patient is compliant with eDiary completion; that is, they have completed the eDiary questions on at least 5 days each week during the 14 calendar days before the start of the Treatment Period.
5. Patient is compliant with continuing any current PPI (if using) during the 14 calendar days before the start of the Treatment Period. Patients are considered compliant if, as reported in the daily eDiary, they continued taking their current PPI (if using) on at least 5 days each week during the 14 calendar days before the start of the Treatment Period.

   4.2 EXCLUSION CRITERIA 1. Age ≥ 65 years 2. Patient is not fluent and literate in English. 3. Pregnant (or plan to be) and nursing mothers 4. Women of child-bearing potential not willing to comply with contraceptive requirements during the study treatment and for 1 week following the last dose of study drug.

   o Definition of women of child-bearing potential

   Non-post-menopausal female, who has not had a bilateral oophorectomy or medically documented ovarian failure. A subject may be considered to be post-menopausal when there is either:

   - twelve (12) months of spontaneous amenorrhea or;

   - six (6) months of spontaneous amenorrhea with serum FSH levels > 40 mIU/mL or;

   - six (6) weeks postsurgical bilateral oophorectomy with or without hysterectomy.

   A female who has had a tubal ligation sterilization or hysterectomy would not be considered to be of reproductive potential unless participating in activities of reproductive potential other than heterosexual intercourse (e.g., egg donation, participation in in vitro fertilization).
   * Contraceptive requirements Fosamprenavir may decrease the effectiveness of combined hormonal contraception through significant CYP3A4 induction of estrogen. If subjects' preferred choice of contraception is combined hormonal contraception, subjects must also agree to use a second method of contraception (condom + spermicide) during study drug treatment.

   Other acceptable highly effective forms of contraception include:
   * Medroxyprogesterone acetate injectable
   * Intrauterine Device
   * Female Sterilization
   * Male Sterilization 4. Currently being treated with another investigational medical device and/or drug 5. A history of gastric or esophageal surgery 6. Gastrointestinal disease that might interfere symptom questionnaire, e.g. inflammatory bowel syndrome 7. A history of laryngeal or neck surgery including thyroidectomy and laryngomicroscopic surgery 8. Suspected esophageal cancer 9. Nasopharyngeal cancer 10. Previously undergone anti-reflux surgery 11. Polypharmacy (five or more concurrent medications due to comorbidities) 12. Any contraindications to FOS including the following:

a. Patients with previously demonstrated clinically significant hypersensitivity (e.g., Stevens-Johnson syndrome) to any of the components of this product or to amprenavir.

b. Patients taking any drugs that are highly dependent on cytochrome P450 (CYP)3A4 for clearance and for which elevated plasma concentrations are associated with serious and/or life-threatening events. Specifically i. Alpha 1-adrenoreceptor antagonist: Alfuzosin ii. Antimycobacterial: Rifampin iii. Antipsychotic: pimozide iv. Ergot derivatives: Dihydroergotamine, ergonovine, ergotamine, methylergonovine v. GI motility agent: Cisapride vi. Herbal product: St. John's wort ( Hypericum perforatum) vii. Lipid modifying agents: Lomitapide, lovastatin, simvastatin viii. Non-nucleoside reverse transcriptase inhibitor: Delavirdine ix. PDE5 inhibitor: Sildenafil (Revatio) x. Sedative/hypnotics: Midazolam, triazolam 13. Patients not willing to avoid eating grapefruit and Seville oranges for five days prior to the first day of dosing study drug through the final study visit.

14. Patients taking any of the prohibited medications or foods listed in Section 5.6.3 15. Anticipated poor understanding or compliance of the study protocol 16. History of hepatic impairment 17. Sulfa Allergy 18. Hemophilia 19. Active tuberculosis (TB) or history of active TB. 20. History of latent TB (e.g., positive QuantiFERON-TB test) without history of active TB unless the subject has completed a documented course of prophylactic treatment.

21. History of human immunodeficiency virus (HIV) infection or positive for HIV 22. . Patients positive for hepatitis (Seropositive for hepatitis B surface antigen [HBsAg] or Hepatitis C virus [HCV] RNA positive) or taking HCV protease inhibitors such as boceprevir, simeprevir and paritaprevir 23. Not willing to refrain from taking biotin containing supplement for at least 12 hours before Visit 1.

24. Patient has an acute or chronic condition that, in the Investigator's opinion, would limit the patient's ability to complete or participate in this clinical study.

25. Additionally, subjects without the following will be excluded:

1. Ownership of an electronic with access to internet websites and email required to conduct the DRSD, PGI-S, and PGI-C
2. Internet access
3. A valid email address for notifications

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 104 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in Reflux Symptom Index (RSI) | Baseline to 12-week post-treatment.
  The absolute change from baseline (i.e., Pretreatment) in symptom severity as indicated by RSI Score over time, with the primary treatment comparison at Week 12 (End of Treatment Visit)
Change in Daily Symptom Reflux Diary (DRSD) | Baseline to 12-week post-treatment.
  The absolute change from baseline (i.e., Pretreatment) in symptom severity as indicated by Weekly Total DRSD Score (WTDS) over time, with the primary treatment comparison at Week 12 (End of Treatment Visit)

OTHER OUTCOMES:
Change in Reflux Finding (RFS) | Baseline to 12-week post-treatment.
  The absolute change from baseline in endoscopic signs severity as indicated by Reflux Finding Score (RFS) over time, with the primary treatment comparison at Week 12
Change in Reflux Symptom Scale (RSS). | Baseline to 12-week post-treatment.
  The absolute change from baseline in symptom severity as indicated by Reflux Symptom Score (RSS) over time, with the primary treatment comparison at Week 12
Change in Reflux Sign Assessment (RSA) | Baseline to 12-week post-treatment.
  The absolute change from baseline in endoscopic signs severity as indicated by Reflux Sign Assessment (RSA) score over time, with the primary treatment comparison at Week 12
Change in Voice Handicap Index 10 (VHI-10) | Baseline to 12-week post-treatment.
  The absolute change from baseline in symptom severity as indicated by Voice Handicap Index-10 (VHI-10) score over time, with the primary treatment comparison at Week 12
Change in Reflux Symptom Index (RSI) | Baseline to week 4 post-treatment.
  The absolute change from baseline in symptom severity as indicated by RSI score over time, (up to Week 4), with the primary treatment comparison at Week 4

CONTACTS AND LOCATIONS:
Locations (1):
- Froedtert Hospital, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No